CLINICAL TRIAL: NCT06032520
Title: The Effectiveness of Forensic Outpatient Systemic Therapy: a Multiple Case Experimental Design
Acronym: FAST
Status: Recruiting | Type: Observational
Sponsor: Utrecht University (Other)
Collaborators: De Waag (Unknown)
Responsible Party: Principal Investigator, Marjolein van Cappellen, PhD Student, Utrecht University
Other Study IDs: 60-63600-98-1138a
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Conduct Disorder; Antisocial Behavior; Aggression; Behavioral Disorder
Keywords: Multiple Case Experimental Design; Forensic Outpatient Systemic Therapy; Antisocial Behavior; Aggression; Mediation; Effectiveness
MeSH Terms: conditions — Conduct Disorder; Antisocial Personality Disorder; Aggression; Mental Disorders; Negotiating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Forensic Outpatient Systemic Therapy (FAST): FAST is a promising treatment for juveniles showing severe antisocial behavior, including aggression, (domestic) violence, and delinquent behavior. FAST has a flexible intensity and length, addresses individual and systemic risk and protective factors, and is responsive to the abilities of the client (system), intervention characteristics all considered crucial for effective treatment.
  Interventions: Behavioral: FAST

INTERVENTIONS:
Behavioral: FAST — FAST includes around 3 hours of face-to-face direct treatment time weekly and consists of a maximum of 10% online direct treatment time (i.e., treatment via phone, video-calling or texting). The treatment stage of FAST lasts five to nine months depending on the individual goals of the juvenile and the caregiver(s) and is followed by a period of aftercare.
  Other Names: Forensic Outpatient Systemic Therapy; Forensische Ambulante Systeem Therapie

SUMMARY:
The purpose of this study is to investigate the effectiveness and mediators of Forensic Outpatient Systemic Therapy (FAST).

DETAILED DESCRIPTION:
Forensic Outpatient Systemic Therapy (in Dutch: Forensische Ambulante Systeem Therapie; FAST) is a promising treatment for juveniles showing severe antisocial behavior, including aggression, (domestic) violence, and delinquent behavior. FAST has a flexible intensity and length, addresses individual and systemic risk and protective factors, and is responsive to the abilities of the client (system), intervention characteristics all considered crucial for effective treatment. The current study will investigate whether FAST is effective in reducing aggression of the juvenile, in reaching client formulated subgoals, and in improving family functioning (i.e., reducing juvenile-caregiver conflict and increasing caregiver responsiveness). In addition, processes of change will be examined, as well as mediation by reaching client formulated subgoals and improved family functioning. A Multiple Case Experimental Design (MCED) with an ABC design will be performed (A = baseline, B = intervention, and C = follow-up). Juveniles with primary aggression and/or anger problems (N = 15) and their caregiver(s) will be recruited.

ELIGIBILITY:
FAST therapists determine whether clients meet inclusion and exclusion criteria of FAST during the standard intake procedure of FAST. The FAST inclusion criteria are:

1. Juvenile has an estimated IQ-score of 80 or higher and/or sufficient adaptive skills to benefit from FAST;
2. Juvenile is aged 12 to 21 years old at the start of the intervention;
3. Juvenile exhibits externalizing behavior resulting in problems in at least two life areas (family, school, or leisure time), determined by clinical impressions based on information from intake and/or referrer information;
4. Juvenile has a medium to high recidivism risk, measured by the Risk Assessment Instrument for Outpatient Forensic Mental Health Care Youth (RAF GGZ Youth);
5. Presence of juvenile-caregiver relationship problems, measured by the RAF GGZ Youth;
6. Juvenile has a diagnosis of a DSM-5 behavioral disorder, which is determined using a new diagnostic process or case file analysis;
7. Juvenile and caregiver(s) cannot be motivated to follow treatment at the treatment site after multiple attempts by the therapist;
8. Juvenile resides with their caregiver(s) or is expected to return to residing with their caregiver(s) within the first two months of FAST.

The FAST exclusion criteria are:

1. Juvenile exhibits severe psychiatric symptoms requiring admission;
2. Problem behavior of the juvenile is caused primarily by substance abuse problems and it is expected that treatment of the substance abuse problems will decrease the problem behavior;
3. The safety of the family members or therapist cannot be sufficiently guaranteed.

To be eligible for participation in this study, one modified study inclusion criterium applies, i.e., the juvenile has primary aggression and/or anger problems (approximately 80% of referred juveniles). In addition, one study exclusion criterium applies, i.e., the juvenile is in secure residential care or confined in a correctional or detention facility at start of the intervention.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes juveniles that will receive FAST. FAST is offered by de Waag, an outpatient forensic mental health care center in the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in Aggression assessed by the Aggressive Behavior scale of the Youth Self Report (YSR) | Twice a week during phase A, up to 5 weeks; every other week during phase B, up to 8 months; weekly during phase C, 6 weeks
  The YSR is a self-reported instrument. The Aggressive Behavior scale contains 19 items assessing aggression. Possible scores range from 1 (never) to 100 (always).
Change in Aggression assessed by the Aggressive Behavior scale of the Child Behavior Checklist (CBCL) | Twice a week during phase A, up to 5 weeks; every other week during phase B, up to 8 months; weekly during phase C, 6 weeks
  The CBCL is a caregiver-reported instrument. The Aggressive Behavior scale contains 19 items assessing aggression. Possible scores range from 1 (never) to 100 (always).
Change in Client Formulated Subgoals assessed by the FAST Goal list | Twice a week during phase A, up to 5 weeks; every other week during phase B, up to 8 months; weekly during phase C, 6 weeks
  The FAST Goal list is a self-report instrument for juveniles and caregivers. It contains 21 items with possible scores ranging from 0 (not true at all) to 100 (definitely true). The FAST Goal lists are used in an idiographic and client-guided approach. The first questionnaire in phase A contains the entire FAST Goal list and a follow-up question asks participants to prioritize their top three FAST goals. In the subsequent measurements, only the items measuring the three prioritized goals are administered. Added to these three items, a fourth item measures whether prioritization or goals have changed. If so, the participant is asked to state their new prioritization or goals, and the questions about the new goals are added in the subsequent measurements.
Change in Juvenile-Caregiver Conflict assessed by the Network of Relationship Inventory (NRI) | T1 (baseline); twice a week during phase A, up to 5 weeks; every other week during phase B, up to 8 months; T2 (post-intervention) up to 9 months; weekly during phase C, 6 weeks
  The NRI is a self-reported instrument for juveniles and caregivers. The NRI contains six items with possible scores ranging from 1 (not at all) to 100 (the most).
Change in Caregiver Responsiveness assessed by the the Responsiveness Scale of the Nijmeegse Parenting Questionnaire (NPQ) | T1 (baseline); twice a week during phase A, up to 5 weeks; every other week during phase B, up to 8 months; T2 (post-intervention) up to 9 months; weekly during phase C, 6 weeks
  The NPQ is a self-reported instrument for juveniles and caregivers. The the Responsiveness Scale contains eight items with possible scores ranging from 1 (completely disagree) to 100 (completely agree).
Change in Additional Criminogenic Needs assessed by individualized items | Twice a week during phase A, up to 5 weeks; every other week during phase B, up to 8 months; weekly during phase C, 6 weeks
  If severe truancy, substance use, contact with deviant peers, or delinquent behavior are reported at T1 but not prioritized in the top three goals, single items will be administered on these problems as well.

SECONDARY OUTCOMES:
Change in Externalizing Behavior assessed by the Youth Self Report (YSR) | T1 (baseline); T2 (post-intervention) up to 9 months
  The YSR is a self-reported instrument. The Externalizing scale contains 30 items assessing aggression and delinquency. Possible scores range from 0 (never) to 2 (often).
Change in Externalizing Behavior assessed with the Child Behavior Checklist (CBCL) | T1 (baseline); T2 (post-intervention) up to 9 months
  The CBCL is a caregiver-reported instrument. The Externalizing scale contains 36 items assessing aggression and delinquency. Possible scores range from 0 (never) to 2 (often).
Change in Delinquency assessed with the Self-Report Delinquent Behavior (SDB) | T1 (baseline); T2 (post-intervention) up to 9 months
  The SDB is a self-reported instrument, assessing how many times the juvenile has done certain (rule-breaking) things in the past year. The SDB contains 30 items.
Percentage of Participants with Out of Home Placement assessed using File Analysis | T1 (baseline); T2 (post-intervention) up to 9 months
  A participant is viewed as being placed out of home when they do not reside with their primary family, either temporarily or permanently, and either voluntarily or involuntarily. Out of home placement is registered by therapists during treatment as part of the standard FAST procedure.
Percentage of Participants with Out of Home Placement assessed using an Out of Home Placement Questionnaire | T2 (post-intervention) up to 9 months
  A participant is viewed as being placed out of home when they do not reside with their primary family, either temporarily or permanently, and either voluntarily or involuntarily. Out of home placement will be assessed using a questionnaire measuring living situation, which is filled in by juveniles and caregivers. The questionnaire contains one item assessing where the juvenile lives most days of the week.
Change in Recidivism Risk assessed with the RAF GGZ Youth | T1 (baseline); T2 (post-intervention) up to 9 months
  The RAF GGZ Youth is an extensive risk assessment instrument and includes items measuring recidivism risk. The RAF GGZ Youth is filled in by the therapist as part of the standard FAST procedure. Possible scores range from 1 (low) to 5 (high).
Change in Substance Use assessed with the Peilstation Middelengebruik | T1 (baseline); T2 (post-intervention) up to 9 months
  Peilstation Middelengebruik is a self-reported instrument. It contains five items assessing frequency and intensity of substance use.
Change in Substance Use assessed with the RAF GGZ Youth | T1 (baseline); T2 (post-intervention) up to 9 months
  The RAF GGZ Youth is an extensive risk assessment instrument and includes items measuring substance use. The RAF GGZ Youth is filled in by the therapist as part of the standard FAST procedure.
Change in Substance Use assessed with the FAST Goal list | T1 (baseline); T2 (post-intervention) up to 9 months
  The FAST Goals List is filled in by juveniles, caregivers, and therapists as part of the standard FAST procedure, and assess the achievement of FAST goals in the past two months. The list includes 1 item on change in substance use. Possible scores range from 1 (not true at all) to 10 (absolutely true).
Change in Contact with Deviant Peers assessed with the Basic Peer Questionnaire (BPQ) | T1 (baseline); T2 (post-intervention) up to 9 months
  The BPQ is a self-reported instrument with 13 items. Possible scores differ per question, for instance measuring amount of friends, or 0 (never) to 4 (5 times or more).
Change in Social Support assessed by the Parental Support Questionnaire (PSQ) | T1 (baseline); T2 (post-intervention) up to 9 months
  The PSQ is a caregiver self-reported instrument and contains 15 items. Possible scores range from 0 (no) to 1 (yes), and 1 (unsatisfied) to 5 (satisfied).
Change in Caregiver-Adolescent Relationship Quality assessed by the Inventory of Parent and Peer Attachment (IPPA) | T1 (baseline); T2 (post-intervention) up to 9 months
  The IPPA is a juvenile self-reported instrument and contains 12 items per caregiver. Possible scores range from
  1 (almost never) to 4 (almost always).
Change in Caregiver-Adolescent Relationship Quality assessed by the Nijmeegse Parenting Stress Index (NPSI) | T1 (baseline); T2 (post-intervention) up to 9 months
  The NPSI is a caregiver self-reported instrument and contains nine items. Possible scores range from 1 (not applicable at all) to 6 (completely applicable).
Change in Caregiver Consistency assessed by the Consistency Scale of the Parenting Dimensions Inventory (PDI) | T1 (baseline); T2 (post-intervention) up to 9 months
  The PDI is a juvenile and caregiver self-reported instrument. The Consistency scale contains eight items. Possible scores range from 1 (completely disagree) to 6 (completely agree).
Change in Behavioral Control assessed by the Parenting Practices | T1 (baseline); T2 (post-intervention) up to 9 months
  The Parent Practices is a juvenile and caregiver self-reported instrument and contains six items. Possible scores range from 1 (never) to 5 (always).
Change in Discipline Practices assessed by the Parenting Dimensions Inventory (PDI) | T1 (baseline); T2 (post-intervention) up to 9 months
  The PDI is a juvenile and caregiver self-reported instrument and contains three hypothetical situations with six items each. Possible scores range from 1 (very improbable) to 6 (very probable).
Change in Psychological Control assessed by the Psychological Control Scale Youth Self-Report (PCS-YSR) | T1 (baseline); T2 (post-intervention) up to 9 months
  The PCS-YSR is a self-reported instrument and contains eight items. Possible scores range from 1 (not applicable at all) to 5 (completely applicable).
Change in Caregiver Competence assessed by the Nijmeegse Parenting Stress Index (NPSI) | T1 (baseline); T2 (post-intervention) up to 9 months
  The NPSI is a caregiver self-reported instrument and contains 15 items. Possible scores range from 1 (completely disagree) to 6 (completely agree).
Change in Parental Monitoring assessed by the Parental Monitoring Scale | T1 (baseline); T2 (post-intervention) up to 9 months
  The Parental Monitoring Scale is reported on by juveniles. It contains five items and one additional item measuring parental knowledge about school grades. Possible scores range from 1 (nothing) to 4 (everything).
Change in Cognitive Distortions assessed by the Brief Irrational Thoughts Inventory (BITI) | T1 (baseline); T2 (post-intervention) up to 9 months
  The BITI is a self-reported instrument and is filled in by juveniles as part of the standard FAST procedure. The BITI contains 18 items with possible scores range from 1 (completely disagree) to 6 (completely agree).
Demographics assessed by a Demographic Information Questionnaire | T1 (baseline)
  The Demographic information questionnaire contains items about gender, age, and occupation. The questionnaire contains nine items for juveniles, 19 for caregivers, and eight for therapists.
Primary Diagnosis assessed by Therapist File Search | T1 (baseline)
  The therapist file contains the primary diagnosis of the juvenile.
Change in Personality assessed by the Inventory of Callous-Unemotional Traits (ICU) | T1 (baseline)
  The ICU is reported by juveniles and caregivers and contains 24 items. Possible scores range from 1 (completely untrue) to 4 (always true).
Change in Personality assessed by the Narcissism and Impulse Control scales of the Antisocial Process Screening Device (APSD) | T1 (baseline)
  The APSD is reported by juveniles and caregivers. The scales contain 12 items for juveniles and 16 items for caregivers. Possible scores range from 1 (completely true) to 4 (always true).
Caregiver Psychopathology assessed by the RAF GGZ Youth | T1 (baseline)
  The RAF GGZ Youth is an extensive risk assessment instrument and includes items measuring caregiver psychopathology. The RAF GGZ Youth is filled in by the therapist as part of the standard FAST procedure. Possible scores range from 0 (problems not present) to 2 (problems definitely present).
Treatment Integrity assessed by the FAST Evaluation Forms | T2 (post-intervention) up to 9 months from baseline
  The FAST evaluation forms are filled in by juveniles, caregivers, and therapists as part of the standard FAST procedure. Possible scores range from 0 (no) to 1 (yes), and 1 (very bad, never) to 10 (very good, always).
Treatment Completion assessed by Therapist File Search | T2 (post-intervention) up to 9 months from baseline
  Treatment completion will be assessed by coding whether FAST completion was registered as positive or negative.
Treatment Duration assessed by Therapist File Search | T2 (post-intervention) up to 9 months from baseline
  Treatment duration will be calculated based on the registered direct treatment time by therapists in their appointment agendas. Treatment duration will be measured in weeks.
Treatment Intensity assessed by Therapist File Search | T2 (post-intervention) up to 9 months from baseline
  Treatment intensity will be calculated based on the registered direct treatment time by therapists in their appointment agendas. Treatment intensity will be measured in average hours of direct treatment time per week.
Therapist-Client Alliance assessed by the Relationship with Interventionist | T2 (post-intervention) up to 9 months from baseline
  The Relationship with Interventionist is a juvenile and caregiver self-reported instrument and contains 12 items. Possible scores range from 1 (completely disagree) to 6 (completely agree).
Change in Treatment Motivation assessed by the Treatment Motivation Scales for Forensic Outpatient Treatment (TMS-F) | T1 (baseline); T2 (post-intervention) up to 9 months
  The TMS-F is reported on by juveniles and caregivers and contains 16 items. Possible scores range from 1 (completely disagree) to 5 (completely agree).
Treatment Expectancies assessed by the Parent Expectancies for Therapy Scale (PETS) | T1 (baseline)
  The PETS is a caregiver self-reported instrument and contains seven items. Possible scores range from 1 (completely disagree) to 5 (completely agree).
Treatment Cooperation assessed by the Cooperation Scale | T2 (post-intervention) up to 9 months from baseline
  The Cooperation Scale is reported on by juveniles, caregivers, and therapists and contains five items. Possible scores range from 1 (completely disagree) to 6 (completely agree).

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - de Waag, Utrecht
  - Utrecht University, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
The details on which parts of the data will be shared still have to be discussed.

REFERENCES:
- See also: FAST Intervention Description — https://www.nji.nl/interventies/forensische-ambulante-systeem-therapie-fast